CLINICAL TRIAL: NCT05545150
Title: Volumetric Lumpectomy Specimen Image Visualization for Intraoperatively Directing Cavity Shaves, a Phase II Study (VIVID)
Brief Title: Volumetric Specimen Imager Device for the Intraoperative Imaging of Patients With Breast Carcinoma and Breast Ductal Carcinoma In Situ, The VIVID Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NU 21B01; NCI-2022-02064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00214652; NU 21B01 (Other: Northwestern University); P30CA060553 (NIH); R44CA206801 (NIH)
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Bilateral Breast Carcinoma; Breast Ductal Carcinoma In Situ; Invasive Breast Carcinoma; Multicentric Breast Carcinoma; Prognostic Stage 0 Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (Volumetric Specimen Imager Device) (Experimental): Patients undergo breast conservation surgery (lumpectomy or partial mastectomy) per standard care, and VSI intraoperative imaging is captured on the day of surgery.
  Interventions: Procedure: Intraoperative Imaging; Device: Lumpectomy

INTERVENTIONS:
Procedure: Intraoperative Imaging — Clarix Imaging Volumetric Specimen Imager
Device: Lumpectomy — Per standard of care (SOC)
  Other Names: Lumpectomy of Breast; Partial Mastectomy

SUMMARY:
This clinical trial assesses if the use of a three-dimensional imaging device called the Clarix Imaging Volumetric Specimen Imager (VSI) can help guide and assist surgeons in identifying and removing all positive margins while in the operating room (intraoperative imaging) for patients with breast cancer and breast ductal carcinoma in situ. Breast conservation surgery or lumpectomy is a standard of care (routine) procedure that removes the tumor and a rim of surrounding normal tissue (margins) while leaving as much normal breast tissue as possible. A margin that does not contain tumor cells is called a negative margin and tells the surgeon that the primary tumor has been removed. A positive margin contains tumor cells at or near the edge of the tissue removed. As part of standard of care, surgeons take two-dimensional x-ray images of the tissue that has been removed in the operating room to assess if there is any additional tissue that should be shaved (removed) to get a negative margin. After the surgery is over, the tissue is examined once again by a pathologist in a laboratory to determine if there are any small pieces of tumor left in the margin that were not visible during surgery. If residual tumor is detected in the margin, a reoperation may be required to remove additional tissue until the tumor has been completely removed from the margin. Diagnostic procedures, such as intraoperative volumetric specimen imaging may reduce the rate of reoperation of for patients who previously underwent lumpectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if intraoperative use of the volumetric specimen imager (VSI) device during breast conservation surgery in women with invasive breast cancer and/or ductal carcinoma in situ (DCIS) allows surgeons to accurately identify margin status, such that =<10% of patients have positive margins on final surgical pathology of the main specimen that were unidentified by VSI image interpretation for excision.

SECONDARY OBJECTIVES:

I. To calculate the sensitivity and specificity of VSI-directed shaves compared to the lumpectomy specimen pathology, when VSI device imaging is used intraoperatively to identify close tumor margins for directed cavity shaving in women with invasive breast cancer and/or DCIS who are undergoing breast conservation surgery.

II. To calculate the length of time spent acquiring images with the VSI device, at the time of breast conservation surgery in women with invasive breast cancer and/or DCIS.

III. To calculate the volume of tissue excised in the main lumpectomy specimen and the volume of tissue excised in VSI-directed cavity shaves, when excising tumor margins at the time of breast conservation surgery in women with invasive breast cancer and/or DCIS.

OTHER PRE-SPECIFIED OBJECTIVES:

I. To compare the estimated final positive margin rate for lumpectomy with VSI-directed cavity shaving to the historical final positive margin rate for lumpectomy with standard of care margin assessment, wherein 'positive margin' is defined per published guidelines.

II. To compare the estimated final positive margin rate for lumpectomy with VSI-directed cavity shaving to the historical final positive margin rate for lumpectomy with standard of care margin assessment, wherein 'positive margin' is defined per institutional practice. III. To compare the estimated reoperation rate for patients undergoing lumpectomy with VSI-directed cavity shaving to the historical reoperation rate for patients who previously underwent lumpectomy with standard of care margin assessment.

EXPLORATORY OBJECTIVE:

I. To retrospectively evaluate the sensitivity and specificity of interpretation of shave margin VSI images to determine the feasibility of imaging shaved margins with VSI to further direct cavity shaves.

OUTLINE:

Patients undergo breast conservation surgery (lumpectomy or partial mastectomy) per standard care, and VSI intraoperative imaging is captured on the day of surgery.

After completion of study, patients are followed up for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with invasive breast cancer and/or ductal carcinoma in situ (DCIS) who will be undergoing breast conservation surgery, consisting of a lumpectomy or partial mastectomy procedure
* Patients must be planning and able to undergo breast conservation surgery with planned localization (any localization device is eligible) and intraoperative imaging for the management of invasive breast cancer and/or DCIS.
* Patients must have histologically confirmed invasive breast cancer, ductal carcinoma in situ (DCIS), or invasive breast cancer with a DCIS component.
* The invasive breast cancer and/or DCIS lesion must have been visualized on mammography/ digital breast tomosynthesis (DBT), ultrasound (US), or magnetic resonance imaging (MRI).

  * Note: Patients with mammographically occult lesions are eligible, provided the lesion can be visualized using MRI or US.
* Patients must be women who are >= 18 years of age.

  * NOTE: Males and children under the age of 18 are not included in this study because the treatment paradigms for these groups are aggressive and routinely include mastectomy, whereas the present study is an investigation of breast conservation.
* The patient (or the patient's legally authorized representative if the patient has impaired decision-making capacity) must have the ability to understand and provide voluntary written informed consent to participate in this study, prior to registration.
* Patients who have received neoadjuvant chemotherapy for the treatment of breast cancer are eligible
* Patients with bilateral breast cancer and/or multicentric disease are eligible.

  * Note: For these patients, the VSI device will only be used on a single lesion
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational intervention for this trial are eligible.

Exclusion Criteria:

* Patients undergoing re-excision for invasive breast cancer or DCIS are not eligible
* Patients who are expected to have an excised lumpectomy specimen that is larger than 9 cm x 9 cm x 7 cm are not eligible

  * Note: The specimen size limitation for the VSI device is 9 cm x 9 cm x 7 cm (length x width x height).
* Patients must not have a physical or psychiatric illness, condition, or social circumstance that the investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Positive margins | Up to 2 months after breast conservation surgery
  The primary endpoint of main specimen positive margins identified by volumetric specimen imager (VSI) interpretation and excised intraoperatively is defined as the proportion of patients with at least one main specimen positive margin that was not excised intraoperatively by a VSI-directed shave. A positive margin is defined as ink on tumor (1 or more tumor cells touching the edge of the lumpectomy specimen) for invasive breast cancer and for invasive breast cancer with a ductal carcinoma in situ (DCIS) component; ink within 2 mm of the edge of the lumpectomy specimen for DCIS, and ink within 2 mm of the lumpectomy specimen for DCIS with microinvasion.

SECONDARY OUTCOMES:
Sensitivity and specificity | Up to 2 months after breast conservation surgery
  The secondary endpoint of sensitivity and specificity of VSI-directed shaves will be determined using data from the surgical pathology report. Sensitivity will be calculated as the proportion of margins with pathologically identified tumor within a range of thresholds from 0-2 mm from the specimen edge directed for shaving by VSI interpretation. Specificity will be calculated as the proportion of margins with pathologically identified tumor above a range of thresholds from 0-2 mm from the specimen edge not directed for shaving by VSI interpretation.
Length of time | Up to 2 months after breast conservation surgery
  Length of time spent acquiring images with the VSI device is defined as the intraoperative time elapsed from the time when VSI imaging is started (i.e., capture of first image frame) to the time when VSI image reconstruction is completed (i.e., three-dimensional [3D] reconstruction image ready for viewing), as reported in the VSI device log file.
Volume of tissue excised | Up to 2 months after breast conservation surgery
  The volume of tissue excised in the main lumpectomy specimen and the volume of tissue excised in VSI-directed shaves is defined as the volume of the main lumpectomy specimen and of the VSI directed shave margins.

OTHER OUTCOMES:
Retrospective analysis per published guidelines | Up to 2 months after breast conservation surgery
  To compare the estimated final positive margin rate for lumpectomy with VSI-directed cavity shaving to the historical final positive margin rate for lumpectomy with standard of care margin assessment, wherein 'positive margin' is defined per published guidelines.
Retrospective analysis per institutional practice | Up to 2 months after breast conservation surgery
  To compare the estimated final positive margin rate for lumpectomy with VSI-directed cavity shaving to the historical final positive margin rate for lumpectomy with standard of care margin assessment, wherein 'positive margin' is defined per institutional practice.
Reoperation rate | Up to 2 months after breast conservation surgery
  To compare the estimated reoperation rate for patients undergoing lumpectomy with VSI-directed cavity shaving to the historical reoperation rate for patients who previously underwent lumpectomy with standard of care margin assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Swati A Kulkarni, MD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - The University of Kentucky, Lexington, Kentucky
  - Washington University in St. Louis, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio